CLINICAL TRIAL: NCT07359014
Title: A Multicenter Clinical Study of Novel CD19/BCMA Dual-Targeted CAR-T Cell Therapy for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Novel CD19/BCMA Dual-Targeted CAR-T Cell Therapy for the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Tongji Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Jinhua Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0650
Record Dates: First submitted 2025-12-31; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Relapse Multiple Myeloma
Keywords: CAR-T therapy

STUDY DESIGN:
Intervention Model Description: relapsed/refractory multiple myeloma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dual CD19/BCMA CAR-T treatment (Experimental): R/R multiple myeloma patients will be treated with novel dual CD19/BCMA CAR-T
  Interventions: Other: Dual CD19/BCMA CAR-T

INTERVENTIONS:
Other: Dual CD19/BCMA CAR-T — Novel CD19/BCMA Dual-Targeted CAR-T Cell Therapy

SUMMARY:
This study aims to investigate the efficacy and safety of CD19/BCMA CAR-T cells in treating relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
B Cell Maturation Antigen (BCMA) Chimeric Antigen Receptor T-cell (CAR-T) therapy is currently a crucial treatment for relapsed/refractory multiple myeloma, yet approximately half of patients still experience relapse with limited subsequent treatment options. Recent studies suggest that dual-target CAR-T may offer new hope for relapsed/refractory multiple myeloma. Preliminary studies in this project demonstrate that the independently designed CD19/BCMA CAR-T exhibits potent anti-myeloma activity both in vitro and in tumor-bearing animal models, positioning it as a potential therapeutic strategy for relapsed/refractory multiple myeloma. Therefore, this study aims to investigate the efficacy and safety of CD19/BCMA CAR-T cells in treating relapsed/refractory multiple myeloma in humans, with the goal of providing novel therapeutic approaches for this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/refractory multiple myeloma.
2. Confirmed by immunohistochemistry (IHC) or flow cytometry of bone marrow samples: plasma cell membrane expression of BCMA is positive (≥30%); no requirement for CD19 positivity rate. All sites must centrally submit bone marrow or plasmacytoma biopsy specimens to the lead site's pathology department or bone marrow/liquid specimens to KingMed Diagnostics (third-party laboratory) for BCMA expression verification.
3. Relapsed/refractory patients must meet the following criteria:

   No response or disease progression after 3 cycles of bortezomib (proteasome inhibitor) or lenalidomide therapy No response or disease progression after 3 cycles of prior treatment regimen Interval between last treatment and disease progression >30 days No current indication for hematopoietic stem cell transplantation (HSCT), or patient refusal of HSCT

   Definition of disease progression follows the 2021 International Myeloma Working Group (IMWG) criteria, meeting at least one of the following:

   Serum M protein ≥ 5 g/L Urine M protein ≥ 200 mg/24 h If serum free light chain (FLC) ratio is abnormal, patient FLC level ≥ 100 mg/L Biopsy-confirmed evaluable plasmacytoma Increased myeloplasmacytic percentage ≥25% (absolute increase ≥10%) Myeloplasm cells constitute ≥30% of total bone marrow cells
4. Expected survival >12 weeks;
5. Disease status is evaluable and meets at least one of the following:

   Serum M-protein ≥10 g/L, 24-hour urine M-protein ≥ 200 mg, Serum FLC ≥ 50 mg/L, Plasmacytoma evaluable by imaging or laboratory testing, Bone marrow plasma cell percentage ≥ 30%
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
7. Sufficient venous access for apheresis or venipuncture, with no other contraindications to blood cell separation;
8. white blood cell (WBC) ≥ 1.5 × 10⁹/L; platelet (PLT) ≥ 45 × 10⁹/L.
9. Serum creatinine ≤ 1.5 times the upper limit of normal (ULN).
10. Alanine Aminotransferase (ALT) ≤ 2.5 ULN, Aspartate Aminotransferase (AST) ≤ 2.5 ULN.

All laboratory values within the above ranges must be achieved without ongoing supportive therapy.

Exclusion Criteria:

1. Received systemic therapy such as cyclophosphamide and fludarabine for lymphoma clearance within 2 weeks prior to enrollment or single-cell collection; prior CD19/BCMA CAR-T therapy; or cell or bispecific antibody therapy within 8 weeks prior to treatment.
2. Received bendamustine-containing regimens within 6 months prior to treatment.
3. Hepatitis C virus (HCV) or Human Immunodeficiency Virus (HIV) positive status; any uncontrolled active infection, including active tuberculosis or Hepatitis B virus (HBV) DNA levels ≥1×10³ copies/mL.
4. Active infection within 72 hours prior to treatment initiation; subjects on ongoing prophylactic antibiotics, antifungals, or antivirals are not excluded provided there is no evidence of active infection and the antibiotics are not on the prohibited drug list.
5. Current systemic use of cyclosporine or steroids such as dexamethasone; recent or current use of inhaled steroids is not exclusionary.
6. Renal impairment with serum creatinine >1.5 times the upper limit of normal (ULN).
7. Hepatic impairment with AST and/or ALT >2.5 times ULN and direct bilirubin >1.5 times ULN.
8. Hyponatremia, serum sodium < 125 mmol/L.
9. Baseline serum potassium < 3.5 mmol/L (exclusion not applied if potassium supplementation prior to study enrollment restores levels above this threshold).
10. Pregnant or lactating women.
11. Other serious conditions that may preclude participation in this trial (e.g., central nervous system disorders, severe heart failure, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, gastric ulcer, active autoimmune disease, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | up to 24 weeks
  The incidence of adverse events and abnormal laboratory findings that are "possibly" or "definitely" related to the study treatment, occurring at any time from the start of monitoring until Week 24, including dose-limiting toxicity (DLT).
Primary implant endpoint | up to 2 years
  The survival time of CAR-T cells in vivo is defined as the "engraftment endpoint." PCR detection of CAR-T cell DNA sequences begins 24 hours post-infusion at scheduled follow-up time points and continues until any two consecutive tests yield negative results, at which point the "engraftment endpoint" is recorded.

SECONDARY OUTCOMES:
complete response (CR), very good partial response (VGPR), and partial response (PR) | up to 2 years
  According to the International Myeloma Working Group (IMWG) unified response criteria for multiple myeloma
Overall survival | up to 2 years
  Overall survival
Progression-free survival | up to 2 years
  Progression-free survival
Detection and quantification of CD19/BCMA CAR-T cells | up to 2 years
  Detection and quantification of CD19/BCMA CAR-T cells in blood, bone marrow, and/or tumor tissue
Detection and quantification of circulating soluble BCMA | up to 2 years
  Detection and quantification of circulating soluble BCMA
BCMA expression | Throughout the entire follow-up period，up to 2 years
  Evaluate BCMA expression in plasma cells and tumor cells
minimal residual disease (MRD) | up to 2 years
  Evaluate the minimal residual disease (MRD) required for subjects to achieve a complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Dr., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Xuzhao Zhang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No